CLINICAL TRIAL: NCT01231984
Title: Comparison of Glycemic Control in Obese Subjects With Diabetes Using the BD Ultra-Fine™ Nano 4mm x 32G Pen Needle, and Either the BD Ultra-Fine™ Short 8mm x 31G Pen Needle or the BD Ultra Fine™ 12.7mm x 29G Pen Needle
Brief Title: Comparison of Glycemic Control in Obese Diabetics Using Three Different Pen Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DBC-10-SQUIR05
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: diabetes; obesity; hypoglycemia; hyperglycemia; pen needle
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 mm vs. 8 mm (Experimental): Subjects randomized to this study arm first used either the 4 mm x 32G Pen Needle or the 8mm x 31G Pen Needle for 12 weeks (Period 1), then switched to the alternate pen needle (PN) for another 12 weeks (Period 2). Order of PN use was randomly determined.
  Interventions: Device: 4 mm x 32G Pen Needle; Device: 8mm x 31G Pen Needle
- 4 mm vs. 12.7 mm (Experimental): Subjects randomized to this study arm first used either the 4 mm x 32G Pen Needle or the 12.7mm x 29G Pen Needle (PN) for 12 weeks (Period 1), then switched to the alternate PN for another 12 weeks (Period 2). Order of PN use was randomly determined.
  Interventions: Device: 4 mm x 32G Pen Needle; Device: 12.7mm x 29G Pen Needle

INTERVENTIONS:
Device: 4 mm x 32G Pen Needle — During the 12 week study period, subjects use this pen needle with their own pen device for all daily insulin injections they usually administered themselves with a pen device. Subjects follow their usual insulin regimen and there is no upper limit on total daily insulin dosage or number of injections. Subjects are advised to inject straight in when using the 4mm PN, with no pinch up.
  Other Names: BD Ultra-Fine™ Nano pen needle, Catalog number 320122
Device: 8mm x 31G Pen Needle — During the 12 week study period, subjects will use this pen needle with their own pen device for all daily insulin injections they usually administered themselves with a pen device. Subjects follow their usual insulin regimen and there is no upper limit on total daily insulin dosage or number of injections. Subjects are directed to use pinch-up when injecting in the abdomen or thigh with the 8mm PN, and no pinch-up at other injection sites.
  Other Names: BD Ultra-Fine™ Short pen needle, Catalog number 320109
  Arms: 4 mm vs. 8 mm
Device: 12.7mm x 29G Pen Needle — During the 12 week study period, subjects will use this pen needle with their own pen device for all daily insulin injections they usually administered themselves with a pen device. Subjects follow their usual insulin regimen and there is no upper limit on total daily insulin dosage or number of injections. When using the 12.7mm PN, subjects are instructed to insert either at an angle of 45 degrees, or to pinch up and hold the pen device at a 90 degree angle (straight in).
  Other Names: BD Ultra-Fine™ Original pen needle, BD Catalog Number 328203
  Arms: 4 mm vs. 12.7 mm

SUMMARY:
Anxiety about needles is a concern commonly expressed by diabetics when beginning insulin therapy. A shorter, thinner pen needle that delivers insulin with the safety and efficacy profile of longer pen needles may appeal to many diabetic patients as the shorter needle may be perceived as less intimidating and more comfortable. While pen needles of 4 to 8 mm in length are generally used for insulin injection in patients considered thin or normal weight, longer (12.7 mm) needles are still often prescribed for overweight or obese patients with diabetes. Since skin thickness is nearly constant across a range of body mass index (BMI), a clear rationale exists for the use of shorter needles in obese patients. (Gibney et al., CMRO 2010)

The primary purpose of this study is to evaluate whether the BD Ultra-Fine™ Nano 4mm x 32 Gauge(G) pen needle manufactured by Becton, Dickinson and Company (BD) provides equivalent glucose control (as measured by hemoglobin A1c levels) as the BD Ultra-Fine™ 8mm x 31G and the BD Ultra-Fine™ 12.7mm x 29G pen needles in obese subjects with diabetes.

DETAILED DESCRIPTION:
Each subject's participation is expected to last a total of 7 months and includes a screening visit, a three-week wash-in period (one week with each of the three different size pen needles) followed by two consecutive 12 week study periods. The purpose of the three week wash-in period is to minimize the number of dropouts during the following study periods by ensuring that subjects have experience using each of the three study needles and find them generally acceptable for use during the study.

Only subjects who complete the wash-in period and confirm their agreement to continue participating will be randomized into one of the two study arms. Subjects will be randomly assigned to use the BD Ultra-Fine™ 4mm pen needle and either the BD Ultra-Fine™ 8mm pen needle or the BD Ultra-Fine™ 12.7mm pen needle. The randomization will also specify which of the two study pen needles to be used first. Half of the study subjects will use the BD Ultra-Fine™ 4mm and BD Ultra-Fine™ 8mm pen needles (4mm/8mm arm) and the other half will use the BD Ultra-Fine™ 4mm and the BD Ultra-Fine™ 12.7mm pen needles (4mm/12.7mm arm). At the end of the first 12 week study period subjects will switch to the other assigned pen needle for the second and final study period.

Glycemic control (based on HbA1c concentrations) will be assessed at baseline and at the end of each 12 week study period.

ELIGIBILITY:
Inclusion Criteria:

* Insulin requiring diabetics (type 1 or type 2)
* Using a pen device for self-injection of all diabetes-related medications for at least two months prior to screening.
* 18 to 80 years of age, inclusive.
* Body Mass Index of at least 30 kg/m².
* Hemoglobin A1c from 5.5 to 9.5 percent (%), inclusive.
* Self-monitor blood glucose at least twice per day with a memory blood glucose meter, and willing to do so at least twice per day for the duration of the study
* On a stable diabetes treatment regimen (for example, no change to non-insulin therapies)for at least 2 months prior to screening
* Able to read, write and follow instructions in English or Spanish.

Exclusion Criteria:

* Administer insulin with a pump.
* Currently use a syringe to inject insulin or any other diabetes-related medication.
* Pregnancy.
* History of intravenous drug abuse.
* Current status or history of a medical condition that would contraindicate treatment with the study product or other conditions which, in the opinion of the Investigator, would place the subject at risk or have the potential to confound interpretation of the study results (i.e. recent history of ketoacidosis, hypoglycemic unawareness, etc.)
* Participated in any one of the following clinical studies:

  * BDDC-08-011, 'Comparison of Glycemic Control among Diabetics using the 4mm x 32G BD Pen Needle versus the 8mm x 31G BD Pen Needle and the 5mm x 31G BD Pen Needle'.
  * DBC-10-SQUIR04, 'Evaluation of Glycemic Control and User Acceptability of the BD Ultrafine Nano 4mm x 32G Pen Needle for Injection of Long-Acting or Basal Insulin Doses Above 40 Units'
  * DBC-10-EMRLD01, 'Design Validation of BD 5-bevel Pen Needles (4,5 and 8mm) in Subjects with Diabetes'

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Hirsch, MD, Study Director — BD Medical - Diabetes Care
Locations (10):
- United States (10):
  - AMCR Institute, Inc., Escondido, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Springfield Diabetes and Endocrine Center, Springfield, Illinois
  - International Diabetes Center (IDC), Minneapolis, Minnesota
  - Diabetes and Endocrine Associates, Omaha, Nebraska
  - The Molly Diabetes Center for Adults and Children at Hackensack University Medical Center, Hackensack, New Jersey
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Corporate Lane Internal Medicine and Research Center, Virginia Beach, Virginia

REFERENCES:
- [Background] Gibney MA, Arce CH, Byron KJ, Hirsch LJ. Skin and subcutaneous adipose layer thickness in adults with diabetes at sites used for insulin injections: implications for needle length recommendations. Curr Med Res Opin. 2010 Jun;26(6):1519-30. doi: 10.1185/03007995.2010.481203. PMID 20429833
- [Derived] Bergenstal RM, Strock ES, Peremislov D, Gibney MA, Parvu V, Hirsch LJ. Safety and efficacy of insulin therapy delivered via a 4mm pen needle in obese patients with diabetes. Mayo Clin Proc. 2015 Mar;90(3):329-38. doi: 10.1016/j.mayocp.2014.12.014. Epub 2015 Feb 7. PMID 25662503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 380 subjects were screened from the current diabetic patient population at 10 research centers in the US. Of those, 293 subjects met eligibility criteria and were enrolled in the wash-in period.
Pre-assignment Details: Subjects who successfully completed the wash-in period and agreed to participate were further randomized into one of the study arms. Specifically, 274 of 293 subjects who were enrolled in the wash-in period completed the wash-in period and were randomized into one of the two study arms.
Groups:
- 4 mm First (4 vs.8): Subjects randomized to this sequence used the 4mm PN for the first 12 weeks (Period 1), then switched to the 8 mm PN for the next 12 weeks (Period 2).
- 8 mm First (4 vs.8): Subjects randomized to this sequence used the 8mm PN for the first 12 weeks (Period 1), then switched to the 4 mm PN for the next 12 weeks (Period 2).
- 4 mm First (4 vs.12.7): Subjects randomized to this sequence used the 4mm PN for the first 12 weeks (Period 1), then switched to the 12.7 mm PN for the next 12 weeks (Period 2).
- 12.7 mm First ( 4 vs.12.7): Subjects randomized to this sequence used the 12.7 mm PN for the first 12 weeks (Period 1), then switched to the 4 mm PN for the next 12 weeks (Period 2).
Period: Study Period 1
Arm/Group | 4 mm First (4 vs.8) | 8 mm First (4 vs.8) | 4 mm First (4 vs.12.7) | 12.7 mm First ( 4 vs.12.7)
Started | 69 | 70 | 66 | 69
Completed | 57 | 63 | 59 | 60
Not Completed | 12 | 7 | 7 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Did not continue to meet I/E Criteria | 2 | 2 | 2 | 2
Not completed — Screen Failure | 0 | 0 | 0 | 1
Not completed — Non-compliance with study requirements | 5 | 0 | 2 | 1
Not completed — Protocol Violation | 3 | 4 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1
Period: Study Period 2
Arm/Group | 4 mm First (4 vs.8) | 8 mm First (4 vs.8) | 4 mm First (4 vs.12.7) | 12.7 mm First ( 4 vs.12.7)
Started | 57 | 63 | 59 | 60
Completed | 54 | 61 | 59 | 56
Not Completed | 3 | 2 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 3
Not completed — Did not continue to meet I/E Criteria | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the population of subjects (274) that completed the wash-in period and were randomized into the study arms.
Groups:
- 4 mm vs. 8 mm: Subjects randomized to this study arm first use either the 4mm PN or the 8mm PN for 12 weeks, then switched to the alternate PN for another 12 weeks. Order of PN use is randomly determined.
- 4 mm vs. 12.7 mm: Subjects randomized to this study arm first use either the 4mm PN or the 12.7mm PN for 12 weeks, then switch to the alternate PN for another 12 weeks. Order of PN use is randomly determined.
- Total: Total of all reporting groups
Arm/Group | 4 mm vs. 8 mm | 4 mm vs. 12.7 mm | Total
Number analyzed (Participants) | 139 | 135 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.6) | 55.9 (11.3) | 56.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 132
  Male | 73 | 69 | 142
Region of Enrollment [Number; unit: participants]
  United States | 139 | 135 | 274

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control as Measured by HbA1c (4 mm vs. 8 mm)
Description: Subjects' glycemic control was assessed by comparing hemoglobin A1c (HbA1c) levels measured at the end of each 12 week Study Period (e.g., at Visit 5 or Visit 7) to the HbA1c measured at the start of that Study Period, i.e. the baseline (Visit 3) for Period 1 and the Period 1/2 crossover (Visit 5) for Period 2.
  Analysis included only subjects with HbA1C values at baseline (Visit 3) and at the end of Study Period 1 (Visit 5) and end of Period 2 (Visit 7).
Time Frame: Over each 12 week study period
Population: 115 subjects completed all main study visits. Two subjects were excluded from the 4 vs. 8 primary analysis due to protocol deviations. The total population size evaluated for the primary objective (4 vs. 8) is therefore 113.
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Groups:
- 4 mm First (4 vs. 8): Subjects randomized to this sequence used the 4mm PN for the first 12 weeks (Period 1), then switched to the 8 mm PN for the next 12 weeks (Period 2).
- 8 mm First (4 vs. 8): Subjects randomized to this sequence used the 8mm PN for the first 12 weeks (Period 1), then switched to the 4 mm PN for the next 12 weeks (Period 2).
Arm/Group | 4 mm First (4 vs. 8) | 8 mm First (4 vs. 8)
Number analyzed (Participants) | 54 | 59
HbA1c (%)
  HbA1c at baseline (Visit 3) | 7.59 (0.86) [-0.209 to 0.058] | 7.46 (1.01) [-0.190 to 0.00]
  HbA1c end of Period 1 (Visit 5) | 7.63 (0.92) | 7.59 (1.28)
  HbA1c end of Period 2 (Visit 7) | 7.78 (1.23) | 7.59 (1.23)
Statistical Analysis 1: Comparison: 4 mm First (4 vs. 8) vs 8 mm First (4 vs. 8); General linear models with baseline as a covariate, needle type, period, and randomization sequence as fixed effects, and subject as random effect were fit to the data; Test type: Non-Inferiority or Equivalence — Two one-sided 95% confidence limits for the difference in HbA1c between the 4mm PN and the 8mm PN was calculated. Equivalence limits for HbA1C were defined a-priori as +/- 0.4% units; Two one-sided 95% confidence limits; For equivalence testing, a 95% test is the same as two one-sided 95% confidence limits; Effect of 4mm versus 8mm PN on HbA1c = -0.076, 95% CI 2-sided [-0.209 to 0.058]

2. Secondary Outcome: Glycemic Control as Measured by HbA1c, in High Dose Insulin (at Least One Dose of ≥ 40 Units) Users
Description: Glycemic control was assessed as by difference between the subjects' HbA1c (%) at baseline (randomization, Visit 3) and at the end of each 12 week study period,in the same manner as for the primary outcome measures. The 95% confidence interval for the mean difference in HbA1c values between the 4mm PN and the longer PN will be estimated based on general linear models adjusting for baseline HbA1c.
Time Frame: Subjects were randomly assigned to use the BD Ultra-Fine™ 4mm pen needle for one - 12 week study period and either the BD Ultra-Fine™ 8mm pen needle or the BD Ultra-Fine™ 12.7mm pen needle for one - 12 week study period.
Population: Of the 226 subjects who were considered for the Primary analysis, 107 subjects had at least one dose of insulin that was at least 40 units. The glycemic control of this sub-group of subjects was analyzed as in the Primary Analysis.The same analysis was performed for the high insulin dose subjects, with the two longer PN study arms pooled together.
Measure: Mean (Standard Deviation); unit: HbA1C (%)
Groups:
- 4 mm First: Subjects in this group first used the 4 mm PN for 12 weeks in Period 1, then switched to a longer PN (8 mm or 12 mm PN) for another 12 weeks in Period 2, based on their randomization.
- Longer PN First (8mm or 12.7mm): Subjects in this group first used one of the longer PNs (8 mm or 12 mm PN) for 12 weeks in Period 1, based on the randomization, then switched to the 4mm PN for another 12 weeks in Period 2.
Arm/Group | 4 mm First | Longer PN First (8mm or 12.7mm)
Number analyzed (Participants) | 52 | 55
HbA1C (%)
  HbA1c at Baseline (Visit 3) | 7.77 (0.92) [-0.230 to 0.051] | 7.57 (0.90)
  HbA1c end Period 1 (Visit 5) | 7.76 (1.03) | 7.62 (0.97)
  HbA1c end Period 2 (Visit 7) | 7.98 (1.35) | 7.66 (0.99)
Statistical Analysis 1: Comparison: 4 mm First vs Longer PN First (8mm or 12.7mm); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Two one-sided 95% confidence limits for the difference in HbA1c between the 4 mm PN and the longer PNs (pooled) was calculated. Equivalence limits for HbA1c were defined a-priori as +/- 0.4% units; Two one-sided 95% confidence limits; For equivalence testing, a 95% test is the same as two one-sided 95% confidence limits; Effect of 4mm PN vs. longer PN on HbA1c = -0.090, 95% CI 2-sided [-0.23 to 0.051]

3. Secondary Outcome: Injection Pain Scores (4 mm vs. 8 mm)
Description: At the end of second study period, subjects were asked to rate the level of pain experienced with study period 2 needle compared to the pen needle used in study period 1, using a 150 mm Visual Analog Scale (VAS). The VAS is a measure of the pain perceived with the needle they are using at that point in the study relative to the needle they used in Period 1. The VAS is anchored at the center (0mm) with "as painful" and at each extreme with "much less painful (-75mm) and "much more painful (+75mm); therefore a pain rating < 0 indicates that the Period 2 needle was perceived as less painful than the Period 1 needle.
Time Frame: At the end of Study Period 2
Population: 115 subjects in the 4mm vs. 8 mm study arm completed all main study visits. Two of the 115 subjects were excluded from all primary and secondary analyses due to protocol deviations. The total number of subjects analyzed for perceived pain for this study was therefore 113.
Measure: Mean (Standard Error); unit: mm
Groups:
- 4 mm Among Those in 8mm x 4 mm Arm: Subjects randomized to this study arm first used the 8mm PN for 12 weeks, then switched to the 4mm PN for another 12 weeks.
- 8 mm Among Those in 4mm x 8mm Arm: Subjects randomized to this study arm first used the 4mm PN for 12 weeks, then switched to the 8mm PN for another 12 weeks.
Arm/Group | 4 mm Among Those in 8mm x 4 mm Arm | 8 mm Among Those in 4mm x 8mm Arm
Number analyzed (Participants) | 59 | 54
mm | -31.53 (5.3) [-75 to 75] | -19.17 (4.85) [-75 to 75]
Statistical Analysis 1: Comparison: 4 mm Among Those in 8mm x 4 mm Arm vs 8 mm Among Those in 4mm x 8mm Arm; Subjects rated the level of pain experienced when using the PN assigned for use during Study Period 2 compared to the PN assigned for use in Study Period 1. By placing a mark on a line, whose midpoint(anchor) was designated as 0, and represented "equivalent pain with assigned PNs", ratings on the continuum represented the degree to which the PN used in the second Study Period was less than or greater than the PN used during the first Study Period; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — p< 0.05 was considered statistically significant in this study; Mean Difference (Final Values) = 12.36, 95% CI 1-sided [lower limit 0.37]

4. Secondary Outcome: Injection Pain Scores (4 mm vs. 12 mm)
Description: At the end of second study period, subjects were asked to rate the level of pain experienced with study period 2 needle compared to the pen needle used in study period 1, using a 150 mm Visual Analog Scale (VAS). The VAS is a measure of the pain perceived with the needle they are using at that point in the study relative to the needle they used the previous period. The VAS is anchored at the center (0mm) with "as painful" and at each extreme with "much less painful (-75mm) and "much more painful (+75mm); therefore a negative pain rating means the period 2 needle was perceived as less painful than the period 1 needle.
Time Frame: At the end of Study Period 2
Population: 115 subjects in the 4mm vs. 12 mm study arm completed all main study visits. One of the subjects was excluded from all primary and secondary analyses due to protocol deviations.
Measure: Mean (Standard Error); unit: mm
Groups:
- 4 mm Among Those in 12mm x 4mm Arm: Subjects randomized to this study arm first used the 12mm PN for 12 weeks, then switched to the 4mm PN for another 12 weeks.
- 12 mm Among Those in 4 mm x 12 mm Arm: Subjects randomized to this study arm first used the 4mm PN for 12 weeks, then switched to the 12mm PN for another 12 weeks.
Arm/Group | 4 mm Among Those in 12mm x 4mm Arm | 12 mm Among Those in 4 mm x 12 mm Arm
Number analyzed (Participants) | 56 | 58
mm | -27.72 (5.47) [-75 to 75] | 3.10 (5.01) [-75 to 75]
Statistical Analysis 1: Comparison: 4 mm Among Those in 12mm x 4mm Arm vs 12 mm Among Those in 4 mm x 12 mm Arm; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — p< 0.05 was considered statistically significant in this study; Mean Difference (Final Values) = 30.83, 95% CI 1-sided [lower limit 18.54]

5. Secondary Outcome: Number of Serious, Unexplained Hypoglycemic Events, Reported as Number of Events by Needle.
Description: Subjects were asked to record hypoglycemic events in his/her diary anytime his/her blood glucose (BG) was below 50mg/dL, s/he had signs/symptoms of hypoglycemia, or s/he required medical attention for treatment.
  Hypoglycemia was defined as serious when the subject required the assistance of another person to be treated, or when the hypoglycemic event met the per-protocol definition of a Serious Adverse Event. An unexplained episode was defined as one with no known cause (for example, the subject skipped a meal or exercised vigorously).
Time Frame: During Study Period 1 (12 weeks) and Study Period 2 (12 weeks)
Population: Two hundred seventy-four subjects were randomized into the study. Data from all subjects randomized were included in the analysis of subjects with serious, unexplained hypoglycemic events.
Measure: Number; unit: Adverse Events
Groups:
- 4mm Needle: Number of subjects enrolled who were assigned to use the 4mm PN.
- 8mm Needle: Number of subjects enrolled who were assigned to use the 8mm PN.
- 12.7mm Needle: Number of subjects enrolled who were assigned to use the 12.7mm PN.
Arm/Group | 4mm Needle | 8mm Needle | 12.7mm Needle
Number analyzed (Participants) | 274 | 139 | 135
Adverse Events | 1 | 2 | 0

6. Primary Outcome: Glycemic Control as Measured by HbA1c (4 mm vs. 12.7 mm)
Description: as for outcome 1
Time Frame: Over each 12 week study period
Population: 115 subjects completed all main study visits. Two subjects were excluded from the 4 vs. 12.7 primary analysis due to protocol deviations. The total population size evaluated for this analysis is therefore 113.
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Groups:
- 4 mm First (4 vs. 12.7): Subjects randomized to this sequence used the 4mm PN for the first 12 weeks (Period 1), then switched to the 12.7 mm PN for the next 12 weeks (Period 2).
- 12.7 mm First (4 vs. 12.7): Subjects randomized to this sequence used the 12.7 mm PN for the first 12 weeks (Period 1), then switched to the 4 mm PN for the next 12 weeks (Period 2).
Arm/Group | 4 mm First (4 vs. 12.7) | 12.7 mm First (4 vs. 12.7)
Number analyzed (Participants) | 57 | 56
HbA1c (%)
  HbA1c Baseline (Visit 3) | 7.57 (0.96) | 7.45 (0.88)
  HbA1c end of Period 1 (Visit 5) | 7.58 (1.03) | 7.54 (0.95)
  HbA1c end of Period 2 (Visit 7) | 7.73 (1.18) | 7.51 (0.97)
Statistical Analysis 1: Comparison: 4 mm First (4 vs. 12.7) vs 12.7 mm First (4 vs. 12.7); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Two one-sided 95% confidence limits for the difference in HbA1c between the 4mm PN and the 12.7mm PN was calculated. Equivalence limits for HbA1C were defined a-priori as +/- 0.4% units; Two one-sided 95% confidence limit; For equivalence testing, a 95% test is the same as two one-sided 95% confidence limits; Effect of 4 mm vs.12.7mm PN on HbA1c = -0.095, 95% CI 2-sided [-0.190 to -0.000]

7. Secondary Outcome: Number of Serious, Unexplained Hyperglycemic Events, Reported as Number of Events by Needle.
Description: Subjects were asked to record hyperglycemic events in his/her diary anytime his/her blood glucose (BG) was above 400mg/dL, or s/he required medical attention for treatment for hyperglycemia.
  Hyperglycemia was defined as serious when the subject required the assistance of another person to be treated, or when the hyperglycemic event met the per-protocol definition of a Serious Adverse Event. An unexplained episode was defined as one with no known cause (for example, the subject missed an insulin dose). Subjects were asked to record these events in a diary.
Time Frame: During Study Period 1 (12 weeks) and Study Period 2 (12 weeks)
Population: Two hundred seventy-four subjects were randomized into the study. Data from all subjects randomized were included in the analysis of subjects with serious, unexplained hyperglycemic events.
Measure: Number; unit: Adverse Events
Arm/Group | 4mm Needle | 8mm Needle | 12.7mm Needle
Number analyzed (Participants) | 274 | 139 | 135
Adverse Events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events that occurred during the wash-in period as well as during the two study periods were collected throughout each subject's participation in the study. Total time of participation could have been up to approximately eight months.
Arm/Group | 4mm Needle | 8mm Needle | 12.7mm Needle
Serious Adverse Events (participants affected / at risk) | 9/274 | 1/127 | 7/147
Other Adverse Events (participants affected / at risk) | 91/274 | 36/127 | 29/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4mm Needle (N=274) | 8mm Needle (N=127) | 12.7mm Needle (N=147)
Diabetic Complications Opthalmic (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic Hernias (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric and Gastroenteric Infections (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal and Abdominal Pains (Excl Oral and Throat) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
General Nutritional Disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Heart Failure NEC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic Conditions NEC (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Inner Ear Signs and Symptoms (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Ulceration and Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Limb Fractures and Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Site Specific Injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Neoplasms Malignant (Excl Islet Cell and Carcinoid) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Urinary Abnormalities (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4mm Needle (N=274) | 8mm Needle (N=127) | 12.7mm Needle (N=147)
Hypoglycaemic Conditions NEC (Metabolism and nutrition disorders) | 60 (209) | 25 (91) | 20 (83)
Hyperglycaemic Conditions NEC (Metabolism and nutrition disorders) | 17 (63) | 8 (20) | 7 (30)
Upper Respiratory Tract Infections NEC (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI and Clinical Center will not publish the results pursuant to the Protocol without sponsor review and opportunity to comment on the publication or oral presentation. Abstracts and synopsis of oral presentations must be received by sponsor 30 days, and journal submissions 60 days, prior to submission. The data generated pursuant to the Protocol will be the property of the sponsor and may be used in any manner by the sponsor as it may determine in its sole discretion.